CLINICAL TRIAL: NCT01748773
Title: Safety and Tolerability of Oxaliplatin-Capecitabine-Trastuzumab Combination and Chemoradiotherapy in Operated Patients With HER-2 Positive Gastric or Gastroesophageal Junction Adenocarcinoma: Phase II Study, TOXAG [ML25574]
Brief Title: A Study of the Combination of Oxaliplatin, Capecitabine, and Trastuzumab With Chemoradiotherapy in the Adjuvant Setting in Operated Participants With Human Epidermal Growth Factor Receptor-2 Positive (HER2+) Gastric or Gastroesophageal Junction Cancer
Acronym: TOXAG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25574
Record Dates: First submitted 2012-12-10; First posted 2012-12-13 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Radiation; Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Therapy (Experimental): Participants will receive combination therapy comprising of trastuzumab, oxaliplatin, capecitabine, and radiation.
  Interventions: Drug: Oxaliplatin; Radiation: Radiation; Drug: Capecitabine; Drug: Trastuzumab

INTERVENTIONS:
Drug: Oxaliplatin — Participants will receive oxaliplatin 100 mg/m^2 IV on Day 1 of Cycles 1-3.
Radiation: Radiation — Participants will receive radiotherapy at total dose of 45 Gy divided into 25 doses, 5 treatments per week for 5 weeks starting on Day 1 of Cycle 4.
Drug: Capecitabine — Participants will receive capecitabine 850 mg/m^2 orally twice daily on Days 1-14 of Cycles 1-3 and on 5 days per week during chemoradiotherapy.
Drug: Trastuzumab — Participants will receive trastuzumab 8 mg/kg IV on Day 1 Cycle 1, 6 mg/kg IV on Day 1 of each following 3-week cycle for 12 months (a total of 17 doses).

SUMMARY:
This single-arm, open-label study will evaluate the safety and efficacy of the combination oxaliplatin, capecitabine, and trastuzumab with chemoradiotherapy in the adjuvant setting in participants with curatively resected HER2+ gastric or gastroesophageal junction cancer. Participants will receive trastuzumab 8 milligrams per kilogram (mg/kg) intravenously (IV) on Day 1 of Cycle 1 and 6 mg/kg IV on Day 1 of every following 3-week cycle, with oxaliplatin 100 milligrams per square meter (mg/m^2) IV on Day 1 of Cycles 1-3, and capecitabine 850 mg/m^2 orally twice daily on Days 1-14 of Cycles 1-3 and on 5 days per week during chemoradiotherapy. Radiotherapy will be given at a total dose of 45 gray (Gy) divided into 25 doses on 5 treatment days each week for 5 weeks starting Day 22 of Cycle 3. Anticipated time on study treatment is 1 year plus a 1-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Curatively resected HER2+ gastric or gastroesophageal junction adenocarcinoma; HER2+ status as defined by immunohistochemistry-2 positive or 3 positive with corroborative Fluorescence In Situ Hybridization+ result
* Participants with stages between Stage IB (T1N1M0) and Stage IIIC
* ECOG performance status score equal to or less than (<=) 2 during screening
* Left ventricular ejection fraction equal to or higher than (>=) 55% with acceptable levels of liver and renal functions
* No known contraindication to capecitabine, oxaliplatin, and trastuzumab
* No contraindication for radiotherapy or has not received any previous radiotherapy to the gastric region for any reason

Exclusion Criteria:

* Participants with a malign condition in the last 5 years except squamous cell carcinoma of the skin
* Previous neoadjuvant chemotherapy and/or radiotherapy
* Any disruption in the physical integrity of the upper gastrointestinal tract (except surgical intervention for gastric or gastroesophageal junction carcinoma)
* Known (previously diagnosed and ongoing) malabsorption syndrome
* Active gastrointestinal bleeding
* Participants with Stage IV gastric or gastroesophageal junction adenocarcinoma
* Clinically significant cardiac or cardiovascular disease
* Uncontrolled hypertension
* Participants who have received any investigational anti-cancer treatment or are being treated in a concomitant investigational drug study
* Abnormal laboratory values at screening for serum total bilirubin, alanine aminotransferase or aspartate amino transferase, alkaline phosphatase, absolute neutrophil count, platelet count, and/or hemoglobin
* Known or suspected hypersensitivity against trastuzumab or proteins of rodents
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-01-29 (Actual); Primary Completion 2015-08-21 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to Month 13
Change from Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status Score | From Baseline to Month 13

SECONDARY OUTCOMES:
Percentage of Participants with Disease-Free Survival, Using Response Evaluation Criteria for Solid Tumors (RECIST) | Cycle 1 Day 1 up to tumor relapse or death due to any reason, whichever occurs first (up to 24 months)
Overall Survival | Cycle 1 Day 1 up to death due to any reason (up to 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Turkey (Türkiye) (9):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital; Medical Oncology, Adana
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Ankara
  - Ankara Oncology Hospital; Oncology, Ankara
  - Baskent University Medical Faculty; Internal Medicine, Ankara
  - Bilkent Sehir Hospita; ONKOLOJI, Çankaya/Ankara
  - Gaziantep University Medical Faculty, Medical Oncology Department, Gaziantep
  - Marmara Uni Faculty of Medicine; Medical Oncology, Istanbul
  - Ege Uni Medical Faculty; Oncology Dept, Izmir
  - Necmettin Erbakan University Meram Medical Faculty ; Internal Diseases, Konya

REFERENCES:
- [Derived] Abali H, Yalcin S, Onal HC, Dane F, Oksuzoglu B, Ozdemir N, Mertsoylu H, Artac M, Camci C, Karabulut B, Basal FB, Budakoglu B, Sendur MAN, Goktas B, Ozdener F, Baygul A. A Phase II Study of the Combination of Oxaliplatin, Capecitabine, and Trastuzumab and Chemoradiotherapy in the Adjuvant Setting in Operated Patients With HER2-positive Gastric or Gastroesophageal Junction Cancer (TOXAG Study): A Turkish Oncology Group Study. Am J Clin Oncol. 2021 Jul 1;44(7):301-307. doi: 10.1097/COC.0000000000000825. PMID 33979100